CLINICAL TRIAL: NCT05662423
Title: The Effects of Expressive Writing Following Traumatic Childbirth
Brief Title: Preventing Childbirth-Related PTSD With Expressive Writing
Acronym: CARES
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Sharon Dekel, PhD, Assistant Professor in Psychology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022P003320
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: PTSD (Childbirth-Related)
Keywords: Mother-Infant Bonding; Postpartum Depression; Postpartum PTSD; Expressive Writing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Depression, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Expressive Writing about Childbirth (Active Comparator): Subgroup of participants will write about their recent childbirth.
  Interventions: Behavioral: Expressive Writing about Childbirth
- Neutral Writing (Placebo Comparator): Subgroup of participants will write about neutral daily events.
  Interventions: Behavioral: Neutral Writing

INTERVENTIONS:
Behavioral: Expressive Writing about Childbirth — Participants will write repeatedly about their deepest emotions and thoughts related to their recent childbirth, focusing on the most stressful experiences.
  Arms: Expressive Writing about Childbirth
Behavioral: Neutral Writing — Participants will write repeatedly about neutral daily events/tasks not related to childbirth.
  Arms: Neutral Writing

SUMMARY:
The goal of this clinical trial is to test a brief psychological intervention given to individuals in the first days following childbirth who have experienced a potentially stressful childbirth. The treatment is aimed at preventing post-traumatic stress disorder following childbirth and promoting maternal-infant bonding.

In the days following childbirth, participants will be asked to write about their childbirth experience or a neutral event for three consecutive days, for around 15 minutes each day. Additionally, they will complete a short survey before and after the intervention about their birth experience and mental health. Around 2 months postpartum (with the option of up to around Month 3 PP), participants will take part in mental health and physiological assessments, and in a brief play session with their infant.

DETAILED DESCRIPTION:
Childbirth-related PTSD (CB-PTSD) is a debilitating maternal mental disorder that undermines the well-being of mothers and can interfere with bonding with their infants during an important time of infant development. A significant portion of delivering women, particularly those who have experienced complicated deliveries, are at-risk for developing CB-PTSD. Underrepresented minorities are also at higher risk for CB-PTSD. An estimated 240,000 American women are likely to be affected by CB-PTSD each year.

Currently, there is no recommended intervention for individuals exposed to traumatic childbirth in hospitals in the United States. Immediate postpartum interventions delivered to at-risk women that are low-cost, low-burden, and feasible are lacking. This study will attempt to fill this gap in effective treatment. Evidence shows that expressive writing (EW), or briefly disclosing in writing mainly thoughts and feelings about a highly stressful event, can have positive effects on mental and physical health. Therefore, the investigators will test the therapeutic effects of EW about recent childbirth in women at-risk for CB-PTSD.

ELIGIBILITY:
Inclusion Criteria:

* Women who recently delivered at Massachusetts General Hospital (MGH).
* Women who are at risk for developing CB-PTSD based on their scoring of >16 on the Peritraumatic Distress Inventory (PDI).

Exclusion Criteria:

* Age <18 or >50.
* Stillbirth.
* Down's Syndrome, other serious genetic disorder in the newborn, or serious birth defect (e.g., microcephaly, spina bifida).
* Admission to the neonatal intensive care unit (NICU) for more than 1 week or infant that is not medically healthy.
* Current diagnosable DSM-5 psychotic or bipolar disorder, or current substance abuse disorder.
* Active suicidality (assessed case by case).
* Present substance abuse as indicated in medical records.
* Severe maternal morbidity (assessed case by case).
* General anesthesia.
* Inability to understand the study procedures, risks, and side effects, or to otherwise give informed consent for participation due to neurological or other reasons.
* Inability to understand English.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in the PTSD Checklist for DSM-5 (PCL-5) total score | Pre-Intervention and Post-Intervention (within 1 day of treatment)
  The PCL-5 is the standard self-report measure to assess PTSD symptom severity. It lists the 20 DSM-5 symptoms regarding a specified event (scale: 0-80, higher scores means worse outcome). In this study the event is specified to recent personal childbirth.
Change from baseline in the PTSD Checklist for DSM-5 (PCL-5) total score | Pre-Intervention and Month 2 postpartum (up to around Month 3 PP)
  The PCL-5 is the standard self-report measure to assess PTSD symptom severity. It lists the 20 DSM-5 symptoms regarding a specified event (scale: 0-80, higher scores means worse outcome). In this study the event is specified to recent personal childbirth.
Physiological reactivity as determined from psychophysiologic responses during script-driven traumatic memory recollection of recent childbirth | Month 2 postpartum (up to around Month 3 PP)
  The posterior probability score will be determined for each participant from a composite of psychophysiological responses during script-driven imagery of recent traumatic childbirth (in comparison to baseline) that includes assessments of heart rate response in beats per minute, skin conductance response in microSiemens, and corrugator frontalis facial muscle electromyogram (EMG) responses in microVolts. The responses to each childbirth script will then be compared with a large database of trauma-exposed subjects by means of a discriminant function analysis, which will yield a posterior probability (PrP) score (higher scores means worse outcome). The PrP scores of the two childbirth scripts will be averaged and will serve as a composite measure of physiological responsivity in the analysis.
Clinician-Administered PTSD-5 Scale for DSM 5 (CAPS-5) | Month 2 postpartum (up to around Month 3 PP)
  The CAPS-5 is the gold-standard interview to diagnose PTSD. It yields a categorical measure of diagnosis and a severity score (scale: 0-80, higher scores means worse outcomes).

SECONDARY OUTCOMES:
Change from baseline in the Mother-to-Infant Bonding Scale (MIBS) total score | Pre-Intervention and Post-Intervention (within 1 day of treatment)
  The MIBS is a simply designed short self-report measure for use from day one postpartum, offering one-word descriptors of possible emotions towards the baby to identify early difficulties in bonding (scale: 0-24, higher scores means worse outcome). This will be assessed in relation to recent childbirth.
Change from baseline in the Mother-to-Infant Bonding Scale (MIBS) total score | Pre-Intervention and Month 2 postpartum (up to around Month 3 PP)
  The MIBS is a simply designed short self-report measure for use from day one postpartum, offering one-word descriptors of possible emotions towards the baby to identify early difficulties in bonding (scale: 0-24, higher scores means worse outcome).This will be assessed in relation to recent childbirth.
Maternal Attachment Inventory (MAI) total score | Post-intervention (within 1 day of treatment)
  The MAI self-report asks about maternal feelings toward and perceptions of the infant; it is considered a robust tool to measure problems in mother-baby relationship (scale: 26-104, higher scores means better outcome). This will be assessed in relation to recent childbirth.
Maternal Attachment Inventory (MAI) total score | Month 2 postpartum (up to around Month 3 PP)
  The MAI asks about maternal feelings toward and perceptions of the infant; it is considered a robust tool to measure problems in mother-baby relationship (scale: 26-104, higher scores means better outcome).This will be assessed in relation to recent childbirth.
Change from baseline in the Edinburgh Postnatal Depression Scale (EPDS) total score | Pre-Intervention and Post-Intervention (within 1 day of treatment)
  The EPDS is a brief 10-item self-report measure (scale: 0-30, higher scores means worse outcome). It recommended for assessing for maternal depression in routine obstetrics care in the US.
Change from baseline in the Edinburgh Postnatal Depression Scale (EPDS) total score | Pre-Intervention and Month 2 postpartum (up to around Month 3 PP)
  The EPDS is a brief 10-item self-report measure (scale: 0-30, higher scores means worse outcome). It recommended for assessing for maternal depression in routine obstetrics care in the US.
Change from baseline in the posttraumatic growth inventory (PTG) total score | Pre-Intervention and Post-Intervention (within 1 day of treatment)
  The PTGI is a 21-item self-report measures that in used in research to assess positive change following a specific (potentially traumatic) event in regard to new possibilities, relating to others, personal strength, spiritual change, and appreciation of Life (scale: 0-125, higher scores means better outcome). This will be assessed in relation to recent childbirth.
Change from baseline in the posttraumatic growth inventory (PTG) total score | Pre-Intervention and Month 2 postpartum (up to around Month 3 PP)
  The PTGI is a 21-item self-report measures that in used in research to assess positive change following a specific (potentially traumatic) event in regard to new possibilities, relating to others, personal strength, spiritual change, and appreciation of Life (scale: 0-125, higher scores means better outcome). This will be assessed in relation to recent childbirth.
Behavioral mother-infant bonding as determined by a quantitative observational assessment of mother-infant interaction using the Coding Interactive Behavior (CIB) | Month 2 postpartum (up to around Month 3 PP)
  Mother-infant bonding behavior will be observed during a 5-min free-play session and coded using the well-validated CIB. The CIB is a global rating system that looks at affective states and interactive styles. Using video-recorded material, the CIB is broken down into 33 codes (18 parent, 8 child, and 7 dyad) rated on a 1-5 scale. Meaningful theory-based constructs, for example, maternal sensitivity (higher scores better outcome), will be used in final analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Yildiz PD, Ayers S, Phillips L. The prevalence of posttraumatic stress disorder in pregnancy and after birth: A systematic review and meta-analysis. J Affect Disord. 2017 Jan 15;208:634-645. doi: 10.1016/j.jad.2016.10.009. Epub 2016 Oct 27. PMID 27865585
- [Background] Pennebaker JW. Expressive Writing in Psychological Science. Perspect Psychol Sci. 2018 Mar;13(2):226-229. doi: 10.1177/1745691617707315. Epub 2017 Oct 9. PMID 28992443
- [Background] Pennebaker JW. Putting stress into words: health, linguistic, and therapeutic implications. Behav Res Ther. 1993 Jul;31(6):539-48. doi: 10.1016/0005-7967(93)90105-4. PMID 8347112
- [Background] Dekel S, Thiel F, Dishy G, Ashenfarb AL. Is childbirth-induced PTSD associated with low maternal attachment? Arch Womens Ment Health. 2019 Feb;22(1):119-122. doi: 10.1007/s00737-018-0853-y. Epub 2018 May 21. PMID 29786116
- [Background] Dekel S, Stuebe C, Dishy G. Childbirth Induced Posttraumatic Stress Syndrome: A Systematic Review of Prevalence and Risk Factors. Front Psychol. 2017 Apr 11;8:560. doi: 10.3389/fpsyg.2017.00560. eCollection 2017. PMID 28443054
- [Background] Chan SJ, Thiel F, Kaimal AJ, Pitman RK, Orr SP, Dekel S. Validation of childbirth-related posttraumatic stress disorder using psychophysiological assessment. Am J Obstet Gynecol. 2022 Oct;227(4):656-659. doi: 10.1016/j.ajog.2022.05.051. Epub 2022 May 29. PMID 35640702
- [Background] Dekel S, Ein-Dor T, Dishy GA, Mayopoulos PA. Beyond postpartum depression: posttraumatic stress-depressive response following childbirth. Arch Womens Ment Health. 2020 Aug;23(4):557-564. doi: 10.1007/s00737-019-01006-x. Epub 2019 Oct 25. PMID 31650283
- [Background] Berman Z, Thiel F, Dishy GA, Chan SJ, Dekel S. Maternal psychological growth following childbirth. Arch Womens Ment Health. 2021 Apr;24(2):313-320. doi: 10.1007/s00737-020-01053-9. Epub 2020 Jul 23. PMID 32705348